CLINICAL TRIAL: NCT00564161
Title: VEGF as a Prognostic Factor for White Matter Damage in Preterm Infants
Status: Withdrawn | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 606060-HMO-CTIL; 606060-HMO-CTIL
Record Dates: First submitted 2007-11-25; First posted 2007-11-27 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2007-11

CONDITIONS: Preterm Infants With White Matter Damage; Preterm Infants Developing Normally

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
We hypothesize that misexpression of vascular endothelial growth factor (VEGF) in the Cerebrospinal fluid of preterm infants can be used as a biomarker to predict the risk for developing white matter damage.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants undergoing lumbar puncture.

Exclusion Criteria:

* Preterm with IVH or known infection or meningitis.

Ages: 25 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm infants.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Study Completion 2009-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Talya Dor, MD, Principal Investigator — Hadassah Medical Organization